CLINICAL TRIAL: NCT05497037
Title: A Prospective, Multicenter, Randomized, Double-Blind, Two-Arm, Sham-Controlled, Parallel-Design Trial to Assess the Efficacy and Safety of Carpal Stim for Treating Carpal Tunnel Syndrome
Brief Title: Safety and Efficacy of Carpal Stim in Treating Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GiMer Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTS001
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Control Group (Sham Comparator): Subject receiving fake stimulation (no stimulation but same device procedure with PRF group)
  Interventions: Device: Sham stimulation
- PRF Group (Active Comparator): Subject receiving 500 KHz PRF stimulation for 15 min
  Interventions: Device: PRF stimulation

INTERVENTIONS:
Device: PRF stimulation — One time 500 kHZ stimulation for 15 min
  Arms: PRF Group
Device: Sham stimulation — Sham stimulation for 15 min
  Arms: Sham Control Group

SUMMARY:
The objective of this study is to assess the efficacy and safety of Carpal Stim for pain relief in CTS subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 20 years old during the recruitment phase
2. Clinical diagnosis of CTS：

   1. Diagnosis of CTS was confirmed by Nerve Conduction Velocity (NCV) but not limited to NCV
   2. Symptoms consistent with CTS for at least 3 months and the numerical rating scale (NRS) score ≥ 5 during the recruitment phase
3. Willing to abstain from any other treatment or therapy for CTS throughout the trial except protocol-described medications
4. The subject is willing and able to comply with the procedure and requirements of this trial
5. The participant is able to understand and provide informed consent, and has signed their written informed consent in accordance with IRB requirements

Exclusion Criteria:

1. Wrist fractures or cysts at the CTS affected side
2. Wrist surgery within the past 3 months, especially carpal tunnel release surgery at the CTS affected side
3. Receiving upper limb (including neck) surgery
4. Injections of corticosteroids/cortisone into the wrist or hand within the past 3 months
5. With a past medical history of diabetic polyneuropathy
6. With a past medical history of rheumatoid arthritis
7. With a past medical history of epilepsy
8. Body Mass Index (BMI) > 40 kg/m2
9. Participation in any investigational study in the last 2 weeks or current enrollment in any trial.
10. Active infection at the stimulator contact site during the recruitment phase
11. Pregnant women or diagnosed with postpartum edema in the wrist per investigator's discretion
12. Patients with implanted medical devices that are electronic products, such as implantable cardioverter defibrillators, pacemakers, spinal cord stimulation systems, or spinal cord drug infusion pumps

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness: The responder rate of the PRF group and Sham-Control group | 1 hour after end of stimulation
Safety: Incidence of adverse events (AEs) and serious AEs (SAEs) | Up to 14 days
Safety: Change in Nerve Conduction Velocity 14th day compared to baseline | 14 days
  Median nerve sensory latency time change over 20%

SECONDARY OUTCOMES:
Proportion in responder in treatment and sham-controlled groups | 3, 7, 14 days after end of stimulation
Change in NRS score in treatment and sham-controlled groups compared to baseline | 1hr, 3, 7, 14 days after end of stimulation
Change in PGIC scale in treatment and sham-controlled compared to baseline | 1hr, 3, 7, 14 days after end of stimulation
Change in GSS score in treatment and sham-controlled compared to baseline | 1hr, 3, 7, 14 days after end of stimulation
Change in BCTQ-SSS score in treatment and sham-controlled compared to baseline | 14 days after end of stimulation
Change in BCTQ-FSS score in treatment and sham-controlled compared to baseline | 14 days after end of stimulation

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Hualien Tzu Chi Hospital, Hualien City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Veterans General Hospital-Taipei, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No